CLINICAL TRIAL: NCT01889134
Title: Osteoprotegerin/sRANKL Ratio and Bone Mineral Density in Patients With Primary Hyperparathyroidism Treated With Parathyroidectomy or Alendronate
Brief Title: OPG/Soluble RANKL (sRANKL) and Bone Mineral Density in Primary Hyperparathyroidism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw Medical University (Other)
Collaborators: Ministry of Science and Higher Education, Poland (Other Government)
Responsible Party: Principal Investigator, Jadwiga Szymczak, assistant professor, Wroclaw Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: GR-722/2009; NN 402 309 536 (Other Grant/Funding Number: Ministry of Science and Higher Education, Poland)
Record Dates: First submitted 2013-06-21; First posted 2013-06-28 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2013-06

CONDITIONS: Primary Hyperparathyroidism
Keywords: primary hyperparathyroidism; RANKL; osteoprotegerin; bone mineral density; alendronate; parathyroidectomy
MeSH Terms: conditions — Hyperparathyroidism, Primary | interventions — Alendronate; Parathyroidectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Alendronate (Experimental): Sedron (alendronate) 70 mg taken orally once a week for 12 months
  Interventions: Drug: Sedron (alendronate)
- Parathyroidectomy (Active Comparator): Selective parathyroidectomy
  Interventions: Procedure: Parathyroidectomy
- Control group (No Intervention): No intervention

INTERVENTIONS:
Drug: Sedron (alendronate)
  Other Names: Alendronate
  Arms: Alendronate
Procedure: Parathyroidectomy
  Arms: Parathyroidectomy

SUMMARY:
The purpose of this study is to determine whether osteoprotegerin and RANKL (receptor activator of nuclear factor-κB ligand) are involved in bone remodeling in patients with primary hyperparathyroidism (PHPT), and whether alendronate may be useful in treatment of the patients with PHPT who are not treated with parathyroidectomy.

DETAILED DESCRIPTION:
Study background and rationale

Receptor activator of nuclear factor-κB (RANK), RANK ligand (RANKL) and its decoy receptor osteoprotegerin (OPG) play key roles in regulating bone turnover. They are involved in the mechanism of "crosstalk" between osteoblasts and osteoclasts. After binding with RANK, RANKL induces bone loss, whereas OPG prevents RANKL-RANK interaction and increases bone mass and strength. The expression of RANKL has been found on the surface of many cell types including cells of the osteoblast lineage, osteocytes, activated T cells and vascular endothelial cells. RANK is a cell bound receptor for RANKL. Its expression has been detected mainly on cells of the macrophage/monocytic lineage, including pre-osteoclastic cells. OPG is produced and secreted by many different cell types including osteoblasts and vascular cells. The OPG/RANKL/RANK system is regulated by many hormones and cytokines among which parathormone (PTH) is one of the most important.

Primary hyperparathyroidism (PHPT) is characterized by sustained secretion of PTH from the parathyroid glands which is excessively disproportionate to calcium levels. This leads to enhanced bone turnover, predominantly resorption, resulting in low bone mass, hypercalcemia, hypercalciuria and hypophosphatemia. Successful parathyroidectomy (PTX) reverses these pathological conditions and is the treatment of choice in PHPT. Alternatively, the bone disease in PHPT may be treated pharmacologically by using bisphosphonates which are able to diminish bone turnover. The mechanism by which PTH exerts its effects in bone and the mechanism of bone loss in PHPT in humans have not been fully explained. PHPT with enhanced PTH seems to be a suitable model to observe possible relationships between PTH, OPG and RANKL.

Study objectives

The primary objective of this study is to investigate the serum Osteoprotegerin/sRANKL (soluble RANKL) ratio in patients with primary hyperparathyroidism who will be treated with parathyroidectomy or with alendronate

Secondary objectives are:

* To compare the effect of parathyroidectomy or treatment with alendronate on bone mineral density (BMD);
* To compare the effect of parathyroidectomy or treatment with alendronate on PTH serum concentration and other biochemical indices of PHPT.

Subjects and control group

The subjects (at least 50) will be recruited from among patients diagnosed with primary hyperparathyroidism while hospitalized in the Department of Endocrinology of Wroclaw Medical University. Before including them in the research they will be thoroughly investigated both in terms of the symptoms of PHPT and other diseases, in particular other hormonal disorders, liver and kidney function during hospitalization.

Patients with symptomatic disease or this who meet surgery criteria will be proposed to undergo a selective PTX. Surgery criteria are generally as follows: a serum calcium concentration >1.0 mg/dL above the upper limit of normal, creatinine clearance <60 mL/min, BMD >2.5 standard deviation below standard reference values for sex-matched peak bone mass at any site (T-score <-2.5), age <50 years old.

Patients who underwent previously unsuccessful parathyroidectomy, who do not meet the criteria for surgery or be unsuitable or unwilling undergo PTX will be treated with alendronate.

The control group will consist of generally healthy volunteers (at least 50) corresponding to the age, gender, and body mass index (BMI) of the patients with PHPT. They should not suffer from bone disease or use medications that could affect BMD and PTH or calcium levels. Healthy people will be used as controls because for many examined parameters the standards of concentrations in serum are not established.

All subjects will sign the informed consent form before entering study. Subjects will have the right to withdraw from the study at any time and for any reason without prejudice to their future medical care by the physician or at the institution.

Study protocol

Patients diagnosed with primary hyperparathyroidism will be destined for PTX (as above) or to treatment with alendronate (Sedron 70 mg once a week taken orally) for one year. From PTX group only patients after successful parathyroidectomy will be followed-up during next 12 months of study.

All subjects will have at least 4 visits: before and after month 3, 6 and 12 during treatment with alendronate or after PTX.

BMD at the lumbar spine (LS), femoral neck (FN), distal third (F-D) and ultradistal (F-UD) sites of the forearm, and of the total body (T) will be measured by dual-energy X-ray absorptiometry (DXA) every six months.

Fasting blood samples as well as 24-h urine specimens will be taken before and after 3, 6 and 12 months of study.

In the control group blood, urine and BMD examination such as in the PHPT group will be carried out once.

Serum and urinary solutes (calcium, phosphate, creatinine) PTH and alkaline phosphatase (ALP) will be assayed in fresh samples. Additionally serum samples will be preserved at -70°C before further hormone and cytokine estimations. The laboratory evaluations will include, but not limited to:

* 1,25-dihydroxyvitamin D (1,25(OH)2D)
* 25-hydroxyvitamin D (25(OH)D)
* Alkaline phosphatase (ALP)
* Calcium
* Creatinine
* C-terminal telopeptide of type I collagen (ICTP)
* Interleukin -18
* Interleukin-1 beta
* Interleukin-6
* Osteocalcin (OC)
* Osteoprotegerin (OPG)
* Parathormone (PTH)
* Phosphate
* Soluble RANKL (receptor activator of nuclear factor-κB ligand)
* Total protein
* Transforming growth factor-beta (TGF-β )
* Tumor necrosis factor-alpha (TNF-α)

The accuracy and completeness of data will be verified by comparing registered data with medical records and paper case report forms.

Safety assessments

Safety assessments will be based on:

* clinical adverse events reported by the subject or observed by the Investigator, including physical examination at all study visits;
* abdominal ultrasound examination every six months;
* laboratory evaluation of serum calcium, phosphate, creatinine at every visit;
* serum pregnancy test, if applicable, done at every visit;
* regular telephone contact with study staff.

Treatment compliance

If a patient misses Sedron administration, he should take the drug next day morning and next dose after one week.

Statistical analysis

The data will be analyzed using Statistica 10 (StatSoft Inc.). Categorical data will be presented by absolute and relative frequencies (n and %). Continuous data will be summarized by the mean, median, standard deviation, minimum and maximum. The pairwise deletion will be used for missing data. The statistical significance of differences between paired data will be calculated using Wilcoxon's signed rank test. The Mann-Whitney U test will be used to compare values between different sample groups. Correlation coefficients will be determined using Spearman's rank correlation. The results will be presented as the mean ± standard deviation. Statistical significance is defined as p<0.05

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of primary hyperparathyroidism
* Subjects able and willing to comply with the requirements of the protocol

Exclusion Criteria:

* Other diseases and medications known to interfere with bone or mineral metabolism, especially bisphosphonates used during the two-year period before this study
* Evidence of active malignancy
* Significant renal impairment as indicated by serum creatinine levels above the normalized range for age
* Significant hepatic dysfunction
* Malabsorption syndrome
* Active gastroduodenal ulcers
* Actual or planned pregnancy (in alendronate group females must not be planning to conceive during the two years following the study) or breast-feeding
* The lack of effective non-hormonal contraception in females with child-bearing capability (in alendronate group)

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2009-01; Primary Completion 2012-06 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in osteoprotegerin/sRANKL ratio at month 12 | 12 months

SECONDARY OUTCOMES:
Changes from baseline in bone mineral density values at month 12 | 12 months
Change from baseline in PTH serum concentration at month 12 | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jadwiga W Szymczak, PhD, MD, Principal Investigator — Wroclaw Medical University (Poland)
Locations (1):
- Department of Endocrinology, Diabetology and Isotope Therapy, Wroclaw Medical University, Wroclaw, Poland